CLINICAL TRIAL: NCT07184736
Title: Comparing Active Versus Passive Aspiration in Therapeutic Thoracentesis: Efficacy, Procedure Time, and Patient Safety
Acronym: Thoracentesis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sheikh Zayed Federal Postgraduate Medical Institute (Other)
Responsible Party: Principal Investigator, Talha Mahmud, Professor Dr. Talha Mahmud, Sheikh Zayed Federal Postgraduate Medical Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: TMahmud; No funding (Other: Department of Pulmonology, Shaikh Zayed Hospital, FPGMI Lahore)
Record Dates: First submitted 2025-09-07; First posted 2025-09-22 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Pleural Effusion
Keywords: Pleural Effusion; Thoracentesis; Active Aspiration; Passive Aspiration; Procedural Complications; Gravity Drainage; Manual Aspiration
MeSH Terms: conditions — Pleural Effusion

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Aspiration (Experimental): For the Active Aspiration Group (n=30), fluid was actively aspirated using a syringe and expelled into a collection bag via a 3-way stopcock.
  Interventions: Procedure: Active Manual Syringe Aspiration
- Passive Aspiration (Experimental): In the passive Aspiration Group (n=30), after initial aspiration to confirm needle placement, the syringe was removed, and fluid was allowed to drain passively via gravity into the collection bag.
  Interventions: Procedure: Passive Gravity Drainage

INTERVENTIONS:
Procedure: Active Manual Syringe Aspiration — For the Active Manual Syringe Aspiration, the operator manually withdraws pleural fluid using a syringe attached to a 3-way stopcock and transfusion set. The fluid is then expelled into a collection bag.
  Arms: Active Aspiration
Procedure: Passive Gravity Drainage — In Passive Gravity Drainage, after confirming proper needle placement with initial aspiration, the syringe is detached, and pleural fluid is allowed to drain passively by gravity through the transfusion set into a collection bag.
  Arms: Passive Aspiration

SUMMARY:
This single-blind randomized controlled trial (RCT) aims to compare the efficacy and safety of active manual aspiration versus passive gravity drainage during therapeutic thoracentesis for large symptomatic pleural effusions. A total of 60 eligible patients will be randomized into two equal groups. The active aspiration group will undergo fluid removal using manual syringe suction, while the passive aspiration group will undergo drainage via gravity. The primary outcomes of the study are the total procedure time and the volume of pleural fluid aspirated. Secondary outcomes include patient-reported pain (measured on a Numeric Rating Scale), patient-reported dyspnea (measured by the mMRC scale), the incidence of procedure-related cough, and the reason for procedure termination. The goal of this study is to determine which technique offers a better balance of efficiency and patient comfort.

ELIGIBILITY:
Inclusion Criteria:

* Patients of either gender.
* Aged above 18 years.
* With symptomatic large pleural effusion (either exudative or transudative).
* Requiring therapeutic pleurocentesis.
* Modified Medical Research Council (mMRC) dyspnea scale grade 3-4.

Exclusion Criteria:

* Uncorrected bleeding diathesis.
* Chest wall cellulitis at the intended site of puncture.
* Uncooperative patients.
* Loculated pleural effusion.
* Traumatic hemothorax.
* Empyema thoracis.
* Hydropneumothorax.
* Patients who refused to participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
Volume of Fluid Aspirated | Immediately upon procedure completion (at the time of needle removal) and fluid extraction.
  The total volume of pleural fluid successfully removed during the procedure, measured in milliliters (ml).
Procedure Time for Therapeutic Thoracentesis | Immediately upon procedure completion (at the time of needle removal) and fluid extraction.
  The total duration of the thoracentesis procedure, measured in minutes, from the initial needle insertion until the procedure was terminated. Termination occurred when no more fluid could be drained, the target volume was reached, or due to patient complications like cough or discomfort.

SECONDARY OUTCOMES:
Patient-Reported Pain | Immediately upon procedure completion (at the time of needle removal) and fluid extraction.
  The level of pain experienced by the patient during or immediately after the procedure, measured using the Numeric Rating Scale (NRS-11), an 11-point scale from 0 (no pain) to 10 (worst pain imaginable).
Patient-Reported Dyspnea | Immediately upon procedure completion (at the time of needle removal) and fluid extraction.
  Description: The level of shortness of breath (dyspnea) was measured using the modified Medical Research Council (mMRC) Dyspnea Scale. The mMRC scale is a 5-point grade-based scale (Range: 0 to 4) used to categorize the severity of a patient's disability due to breathlessness. A higher score indicates a worse outcome.
  Grade 0: No breathlessness except with strenuous exercise. Grade 1: Shortness of breath when hurrying on level ground or walking up a slight hill.
  Grade 2: Walks slower than people of the same age on level ground because of breathlessness, or has to stop for breath when walking at own pace on level ground.
  Grade 3: Stops for breath after walking about 100 meters or after a few minutes on level ground.
  Grade 4: Too breathless to leave the house, or breathless when dressing or undressing.
Incidence of Cough | Immediately upon procedure completion (at the time of needle removal) and fluid extraction.
  The occurrence of cough during or at the end of the procedure, recorded as a binary outcome (yes/no).

OTHER OUTCOMES:
Reason for Procedure Termination | Immediately upon procedure completion (at the time of needle removal) and fluid extraction.
  The specific reason for stopping the procedure, categorized as: (1) target fluid volume (1-1.5L) achieved, or (2) terminated early due to complications (e.g., cough, chest discomfort) or spontaneous drainage cessation.

CONTACTS AND LOCATIONS:
Locations (1):
- Sheikh Zayed Hospital, Lahore, Punjab Province, Pakistan